CLINICAL TRIAL: NCT05473741
Title: Risk of Breakthrough Symptoms On Antipsychotic Maintenance Medication When Remitted Patients Are Treated With Long-Acting Injectable Medications
Brief Title: Risk of Breakthrough Symptoms With Long-Acting Injectable Medications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 176/2020
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Schizophrenia; Schizophrenia Relapse
Keywords: Schizophrenia; Relapse; Long-acting injectable antipsychotics; Remission
MeSH Terms: conditions — Schizophrenia; Recurrence | interventions — Paliperidone Palmitate; Risperidone; Aripiprazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Urine drug screens
  2. Plasma antipsychotic levels
  3. Plasma prolactin levels
  4. Hemoglobin A1c
  5. Lipid panel including total cholesterol, triglycerides, HDL cholesterol and LDL cholesterol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SGA-LAI: Outpatients with schizophrenia treated with second generation long-acting injectable antipsychotics whose psychotic symptoms have remitted.
  Interventions: Drug: Second Generation Long-Acting Injectable Antipsychotic Medications

INTERVENTIONS:
Drug: Second Generation Long-Acting Injectable Antipsychotic Medications — Patients who have been stabilized on long-acting injectable formulations of paliperidone palmitate, risperidone and aripiprazole will be followed for 48 weeks to determine the rate of relapse when adherence is established. Blood samples to measure plasma antipsychotic levels and prolactin levels, and urine samples for drug screen will be collected at baseline and at the 24-week and 48-week time points.
  Other Names: paliperidone palmitate, risperidone, aripiprazole

SUMMARY:
This prospective longitudinal cohort study will follow patients with schizophrenia who are treated with second generation long-acting injectable antipsychotic medications (LAIs) for 48 weeks to determine the risk of psychotic symptom relapse when treatment adherence is established. The study is designed to minimize the other factors that have contributed to breakthrough psychotic symptoms in patients treated with LAIs including poor adherence, substance use, concurrent mood disorders, poor treatment response, failed cross-titration, and insufficient dosing. Eligible subjects will undergo a screening visit to document that inclusion criteria are met and those meeting exclusion criteria are excluded. Participants will be assessed every 12 weeks to determine whether they remain in remission or meet criteria for a relapse. More comprehensive assessment will be completed at the beginning of the study (baseline visit), at the 24-week study midpoint and the 48-week study endpoint. Plasma antipsychotic levels will be measured at these three study time points to investigate associations between plasma levels and remission/relapse status as well as side effects. Plasma prolactin will also be measured to assess the association with sexual side effects. Hemoglobin A1c and measures of total cholesterol, triglycerides, HDL cholesterol and LDL cholesterol will be obtained to assess the effects of SGA LAIs on these measures.

DETAILED DESCRIPTION:
Rationale and Study Objectives In this study, we aim to determine the likelihood that relapse of psychosis will occur when patients with schizophrenia who have experienced a remission of their psychotic symptoms are adherent to treatment with a second generation antipsychotic (SGA) LAI on which they have been stable at a therapeutic dose for at least three months.

Primary objective:

1. To estimate the rate of psychotic relapse in patients with schizophrenia whose psychotic symptoms have remitted and who are adherent with second generation LAIs for maintenance treatment.

Secondary objectives:

1. To determine whether the risk of psychotic relapse is associated with antipsychotic plasma levels in patients treated with second generation LAIs.

Study design:

This prospective longitudinal cohort study will follow patients with schizophrenia who are treated with the second generation LAIs (paliperidone palmitate, risperidone or aripiprazole) for 48 weeks to determine the risk of psychotic symptom relapse when treatment adherence is established. The study is designed to minimize the other factors that have contributed to breakthrough psychotic symptoms in patients treated with LAIs including poor adherence, concurrent mood disorders, poor treatment response, failed cross-titration, and insufficient dosing.

Laboratory tests:

The following laboratory tests will be carried out at the baseline visit, 24-week visit and 48-week visit:

1. Urine drug screen - to document use of cannabis and other common recreational drugs. This will allow us to determine whether substance use is associated with the risk of relapse in remitted patients with established adherence to LAIs.
2. Plasma antipsychotic levels - to determine whether trough (pre-injection) plasma levels are associated with risk of relapse and medication side effects
3. Plasma prolactin - to determine whether the incidence and severity of sexual dysfunction is associated with antipsychotic plasma levels

   The following laboratory tests will be carried out at the baseline visit and 48-week visit:
4. Hemoglobin A1c - to determine the effects of LAIs on blood sugar levels
5. Lipid panel - to determine the effects of LAIs on total cholesterol, triglycerides, HDL cholesterol and LDL cholesterol

The target population is individuals diagnosed with schizophrenia whose psychotic symptoms have remitted and are receiving outpatient care at the Centre for Addiction and Mental Health (CAMH) in Toronto, Ontario, Canada. Patients who have been stabilized on long-acting injectable forms of either paliperidone palmitate, risperidone or aripiprazole with be invited to participate in this study.

Participants will be recruited from CAMH outpatient treatment teams in Toronto, Ontario, Canada, that provide follow-up to individuals diagnosed with schizophrenia including:

1. Downtown Central Flexible Assertive Community Treatment (DC-FACT)
2. Downtown West Flexible Assertive Community Treatment (DW-FACT)
3. Downtown East Flexible Assertive Community Treatment (DE-FACT)
4. Slaight Centre Early Intervention Service (SCEIS)
5. Forensic Outpatient Program for Schizophrenia (FOPS)
6. Psychosis Coordinated Care Service (PCCS)
7. General Psychosis Service (GPS)

All outpatients of the above clinics who are receiving treatment with LAI paliperidone, risperidone, or aripiprazole will be invited to participate in this study if they are considered to meet inclusion criteria and do not meet any of the exclusion criteria listed below. A screening visit will be scheduled for potential participants who express interest in the study. The study and procedures involved with be explained to eligible participants and informed consent will be obtained for study participation by the study research coordinator or research assistant. A baseline visit will then be scheduled.

Study Duration:

The study duration will be 48 weeks rather than 52 weeks as participants treated with LAIs are most commonly administered medication at intervals of two, three, four or twelve weeks. Each of these intervals would fit with major assessments as 24 weeks (study mid-point) and 48 weeks (study end-point).

Study Visit:

At the screening visit, the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) will be administered to determine if the subject meets criteria for schizophrenia and that they do not meet diagnoses that would exclude them from study participation. Screening for other exclusion criteria including medical disorders, concomitant medications, and suicide attempts or hospitalizations in the past 3 months, will be completed at this visit. Subjects who do not meet inclusion criteria or who meet exclusion criteria will be informed and will not participate in further assessments.

Following the Screening visit, all subjects will be assessed at the following time points: Baseline, 12-week, 24-week, 36-week and 48-week visits, with more comprehensive assessments carried out at baseline, 24 weeks and 48 weeks. The following laboratory tests will be carried out at the baseline visit, 24-week visit and 48-week visit: urine drug screen, plasma antipsychotic levels, plasma prolactin. Height will be collected at baseline and weight and waist circumference will be collected at these time points. Hemoglobin A1c and a lipid panel will be obtained at baseline and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 Schizophrenia
* Age 18-65 years
* On SGA LAI: paliperidone palmitate (4-week or 12-week formulations), risperidone or aripiprazole
* Receiving LAI injections through clinical services based at CAMH
* History of improvement in psychotic symptoms with antipsychotic medication as evidenced by a rating of mild or less on the Clinical Global Impression - Severity (CGI-S) for Positive symptoms
* Demonstrated adherence to LAIs defined as not having received any injections more that 7 days past its due date in the past 3 months
* On stable dose of LAI for 3 months or longer
* Capable of providing informed consent for participation in this study

Exclusion Criteria:

* Current DSM-5 major depressive episode or manic episode
* Receiving any oral antipsychotic medication in the past 3 months
* History of organic brain disease (e.g. cerebrovascular accident, Huntington's Disease, Parkinson's Disease, epilepsy, etc.)
* History of untreated or unstable medical illness (e.g. thyroid disease, cancer)
* History of electroconvulsive therapy (ECT) in the past year
* History of suicide attempt in the past 3 months
* History of psychiatric hospitalization in the past 3 months
* Inability to read and communicate in English

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population is individuals diagnosed with schizophrenia whose psychotic symptoms have remitted and are receiving outpatient care at the Centre for Addiction and Mental Health (CAMH) in Toronto, Ontario, Canada. Patients who have been stabilized on long-acting injectable forms of either paliperidone palmitate, risperidone or aripiprazole with be invited to participate in this study. Participants will be recruited from seven CAMH outpatient treatment clinics that provide follow-up to individuals diagnosed with schizophrenia.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impressions Schizophrenia Scale (CGI-SCH) - Positive Symptoms Change subscale | Assessed at 12 weeks, 24 weeks, 36 weeks and 48 weeks
  Subjects will be considered to have relapsed during the study if they are assessed as having a change score of 6 ("much worse") or 7 ("very much worse") on the Clinical Global Impressions Schizophrenia Scale (CGI-SCH) - Positive Symptoms Change subscale (Haro et al., 2003). The minimum score on this scale is "1" - "Very much improved" and the maximum score is "7" - "Very much worse". A higher score means a worse outcome.

SECONDARY OUTCOMES:
Clinical Global Impression Schizophrenia scale | Assessed at 24 weeks and 48 weeks
  Clinical Global Impression Schizophrenia scale (CGI-SCH) (Haro et al., 2003) The minimum score is "1" - "Normal, not ill" and the maximum score is "7" - "Among the most severely ill". A higher score means a worse outcome.
Brief Psychiatric Rating Scale | Assessed at 24 weeks and 48 weeks
  Brief Psychiatric Rating Scale (BPRS) (Overall and Gorham, 1962) This scale measures psychiatric symptoms on a scale from 1-7, where 1 is the least severe and 7 is the most severe. The 24 signifies that it is the longer version of the assessment which includes 24 questions. The minimum score is 24 and the maximum score is 168. A higher score means more severe symptoms/ worse outcome.
Calgary Depression Scale | Assessed at 24 weeks and 48 weeks
  Calgary Depression Scale (CDS) (Addington et al., 1993) This scale is a nine-item structured interview that assesses the level of depression in people with schizophrenia. Items are measured on a 4-point Likert-scale from "0" to "3" where higher ratings indicate more depressive symptoms and a worse outcome. The minimum total score for the scale is "0" and the maximum score is "27" with higher scores indicating more severe depressive symptoms.
VAGUS Insight Into Psychosis Scale | Assessed at 24 weeks and 48 weeks
  VAGUS Insight Into Psychosis Scale (Gerretsen et al., 2014) The VAGUS is a 10-item self-report scale that uses 10-point Likert scales to capture subtle changes in degree of insight into illness. The minimum score is 0 and the maximum score is 10. Higher scores reflect better insight and lower scores indicate poorer insight.
Personal and Social Performance Scale | Assessed at 24 weeks and 48 weeks
  Personal and Social Performance Scale (PSP) (Morosini et al., 2000) This scale assesses a patient's degree of impairment in four domains. Each domain is rated on a six-point scale from absent to very severe. Using the ratings on the four sub-dimensions, one total score on a 100-point scale is created, where 100 is no impairment and 0 is the most severely impaired.
Satisfaction with Life Scale | Assessed at 24 weeks and 48 weeks
  Satisfaction with Life Scale (SWLS) (Diener et al., 1985) This is a 5-item instrument designed to measure global cognitive judgments of satisfaction with one's life. Each item is rated from "0" to "7" with total scores ranging from "0" to "35". Higher scores indicate better outcomes.
Single-Item Happiness Questionnaire | Assessed at 24 weeks and 48 weeks
  Single-Item Happiness Questionnaire (SIQ) (Abdel-Khalek, 2006) This scale involves answering a single question with ratings ranging from "0" to "10" with higher scores indicating better outcomes/greater happiness.
Quality of Life Scale | Assessed at 24 weeks and 48 weeks
  Quality of Life Scale (QLS) (Heintichs et al., 1984) This is a 21-item assessment that evaluates the adequacy of an individual's psychosocial functioning over the past month on 7-point Likert scales (items rate from "0" to "6") with a higher score meaning better functioning. The minimum total score is "0" and the maximum score is "126" with higher scores indicating better outcomes.
UKU Side Effect Rating Scale | Assessed at 24 weeks and 48 weeks
  Udvalg for Kliniske Undersogelser (UKU) Side Effect Rating Scale (Lingjaerde et al., 1987) The scale involves rating 48 side effects on a 4-point scale from "0" to "3" with higher scores indicating more severe side effects.
Subjective Well-Being Under Neuroleptics Scale | Assessed at 24 weeks and 48 weeks
  Subjective Well-Being Under Neuroleptics Scale (SWN) (Naber et al., 2001) This is a self-rated scale consisting of 20 items that are assessed on a 6-point Likert scale. Each item is rated from "1" to "6". The minimum score is 20 and the maximum score is 120. Higher scores indicate better subjective well-being.
Barnes Akathisia Scale | Assessed at 24 weeks and 48 weeks
  Barnes Akathisia Scale (BAS) (Barnes, 1989) This scale is scored on Objective Akathisia, Subjective Awareness of Restlessness and Subjective Distress Related to Restlessness. Each are rated on a 4-point scale from "0" to "3" and are summed to yield a total score ranging from 0 to 9, with 9 being the most severely affected. There is also a Global Clinical Assessment of Akathisia item that is rated from "0" - "Absent" to "5" - "Severe Akathisia".
Arizona Sexual Experiences Scale | Assessed at 24 weeks and 48 weeks
  Arizona Sexual Experiences Scale (ASEX) (McGahuey et al., 2000) This is a five-item rating scale assessing sexual dysfunction with each item rated from "1" to "6". Possible scores range from 5 to 30, with the lower scores indicating better sexual functioning and higher scores indicating worse sexual functioning (i.e. more sexual dysfunction).

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Zipursky, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alphs L, Nasrallah HA, Bossie CA, Fu DJ, Gopal S, Hough D, Turkoz I. Factors associated with relapse in schizophrenia despite adherence to long-acting injectable antipsychotic therapy. Int Clin Psychopharmacol. 2016 Jul;31(4):202-9. doi: 10.1097/YIC.0000000000000125. PMID 26974214
- [Background] Gaebel W, Schreiner A, Bergmans P, de Arce R, Rouillon F, Cordes J, Eriksson L, Smeraldi E. Relapse prevention in schizophrenia and schizoaffective disorder with risperidone long-acting injectable vs quetiapine: results of a long-term, open-label, randomized clinical trial. Neuropsychopharmacology. 2010 Nov;35(12):2367-77. doi: 10.1038/npp.2010.111. Epub 2010 Aug 4. PMID 20686456
- [Background] Gaebel W, Riesbeck M, Wolwer W, Klimke A, Eickhoff M, von Wilmsdorff M, Lemke M, Heuser I, Maier W, Huff W, Schmitt A, Sauer H, Riedel M, Klingberg S, Kopcke W, Ohmann C, Moller HJ; German Study Group on First-Episode Schizophrenia. Relapse prevention in first-episode schizophrenia--maintenance vs intermittent drug treatment with prodrome-based early intervention: results of a randomized controlled trial within the German Research Network on Schizophrenia. J Clin Psychiatry. 2011 Feb;72(2):205-18. doi: 10.4088/JCP.09m05459yel. Epub 2010 Jun 29. PMID 20673559
- [Background] Haro JM, Kamath SA, Ochoa S, Novick D, Rele K, Fargas A, Rodriguez MJ, Rele R, Orta J, Kharbeng A, Araya S, Gervin M, Alonso J, Mavreas V, Lavrentzou E, Liontos N, Gregor K, Jones PB; SOHO Study Group. The Clinical Global Impression-Schizophrenia scale: a simple instrument to measure the diversity of symptoms present in schizophrenia. Acta Psychiatr Scand Suppl. 2003;(416):16-23. doi: 10.1034/j.1600-0447.107.s416.5.x. PMID 12755850
- [Background] Ikai S, Remington G, Suzuki T, Takeuchi H, Tsuboi T, Den R, Hirano J, Tsunoda K, Nishimoto M, Watanabe K, Mimura M, Mamo D, Uchida H. A cross-sectional study of plasma risperidone levels with risperidone long-acting injectable: implications for dopamine D2 receptor occupancy during maintenance treatment in schizophrenia. J Clin Psychiatry. 2012 Aug;73(8):1147-52. doi: 10.4088/JCP.12m07638. PMID 22967779
- [Background] Kapur S, Zipursky R, Jones C, Remington G, Houle S. Relationship between dopamine D(2) occupancy, clinical response, and side effects: a double-blind PET study of first-episode schizophrenia. Am J Psychiatry. 2000 Apr;157(4):514-20. doi: 10.1176/appi.ajp.157.4.514. PMID 10739409
- [Background] Kapur S, Zipursky RB, Remington G. Clinical and theoretical implications of 5-HT2 and D2 receptor occupancy of clozapine, risperidone, and olanzapine in schizophrenia. Am J Psychiatry. 1999 Feb;156(2):286-93. doi: 10.1176/ajp.156.2.286. PMID 9989565
- [Background] Kirson NY, Weiden PJ, Yermakov S, Huang W, Samuelson T, Offord SJ, Greenberg PE, Wong BJ. Efficacy and effectiveness of depot versus oral antipsychotics in schizophrenia: synthesizing results across different research designs. J Clin Psychiatry. 2013 Jun;74(6):568-75. doi: 10.4088/JCP.12r08167. Epub 2013 Apr 19. PMID 23842008
- [Background] Kishimoto T, Hagi K, Nitta M, Leucht S, Olfson M, Kane JM, Correll CU. Effectiveness of Long-Acting Injectable vs Oral Antipsychotics in Patients With Schizophrenia: A Meta-analysis of Prospective and Retrospective Cohort Studies. Schizophr Bull. 2018 Apr 6;44(3):603-619. doi: 10.1093/schbul/sbx090. PMID 29868849
- [Background] Kishimoto T, Nitta M, Borenstein M, Kane JM, Correll CU. Long-acting injectable versus oral antipsychotics in schizophrenia: a systematic review and meta-analysis of mirror-image studies. J Clin Psychiatry. 2013 Oct;74(10):957-65. doi: 10.4088/JCP.13r08440. PMID 24229745
- [Background] Kishimoto T, Robenzadeh A, Leucht C, Leucht S, Watanabe K, Mimura M, Borenstein M, Kane JM, Correll CU. Long-acting injectable vs oral antipsychotics for relapse prevention in schizophrenia: a meta-analysis of randomized trials. Schizophr Bull. 2014 Jan;40(1):192-213. doi: 10.1093/schbul/sbs150. Epub 2012 Dec 17. PMID 23256986
- [Background] Leucht S, Tardy M, Komossa K, Heres S, Kissling W, Salanti G, Davis JM. Antipsychotic drugs versus placebo for relapse prevention in schizophrenia: a systematic review and meta-analysis. Lancet. 2012 Jun 2;379(9831):2063-71. doi: 10.1016/S0140-6736(12)60239-6. Epub 2012 May 3. PMID 22560607
- [Background] Olivares JM, Sermon J, Hemels M, Schreiner A. Definitions and drivers of relapse in patients with schizophrenia: a systematic literature review. Ann Gen Psychiatry. 2013 Oct 23;12(1):32. doi: 10.1186/1744-859X-12-32. PMID 24148707
- [Background] Subotnik KL, Casaus LR, Ventura J, Luo JS, Hellemann GS, Gretchen-Doorly D, Marder S, Nuechterlein KH. Long-Acting Injectable Risperidone for Relapse Prevention and Control of Breakthrough Symptoms After a Recent First Episode of Schizophrenia. A Randomized Clinical Trial. JAMA Psychiatry. 2015 Aug;72(8):822-9. doi: 10.1001/jamapsychiatry.2015.0270. PMID 26107752